CLINICAL TRIAL: NCT07404657
Title: Preliminary Assessment of iCare RETCAD as an Automated Tool for Diabetic Retinopathy Screening
Brief Title: Preliminary Assessment of an Automated Tool for Diabetic Retinopathy Screening
Status: Not yet recruiting | Type: Observational
Sponsor: Centervue SpA (Industry)
Responsible Party: Sponsor
Other Study IDs: RETCAD-PVAL
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Diabetic Retinopathy (DR)
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No

INTERVENTIONS:
Device: automatic analysis of fundus images performed by the software tool based on artificial intelligence — the duration of the intervention is the analysis performed by the software tool based on fundus images acquired

SUMMARY:
This study is being done to evaluate the performance of a software that uses artificial intelligence to analyze photographs of the retina to help detect diabetic retinopathy. The study will also assess the safety of the software in combination with a fundus camera already available on the market. This software analyzes retinal photographs to detect more than mild diabetic retinopathy in adults with diabetes. The results will be compared to expert human evaluations.

ELIGIBILITY:
Inclusion Criteria:

* 22 years old or older
* diabetes or diabetic retinopathy
* understand the study information and able to sign a consent form

Exclusion Criteria:

* cannot tolerate eye imaging tests
* laser treatment or injections
* eye surgery, except for simple cataract surgery
* currently involved in another study
* pregnant
* cannot or do not want to have your eyes dilated
* photodynamic therapy within the last 90 days

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: population attending a primary-care facility with diagnosis of diabetes mellitus and/or past diagnosis of diabetic retinopathy
Sampling Method: Non-Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of subjects whose results provided by the automatic AI-based tool match the reading center grading for the identification of referable diabetic eye disease (more than mild DR). | 1-day visit

SECONDARY OUTCOMES:
percentage of eyes for which the AI-based automatic tool produced a result | 1-day visit